CLINICAL TRIAL: NCT07354438
Title: Assessing the Effect of an Antioxidant-Rich Diet on Metabolic Syndrome Risk Using the Dietary Antioxidant Index
Acronym: AD-MetS-DAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Qaisar Raza, Assistant Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniversityVAS3
Record Dates: First submitted 2025-12-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Syndrome Risk Factors
Keywords: Antioxidants; Dietary antioxidant index; Metabolic Syndrome risk

STUDY DESIGN:
Intervention Model Description: This study uses a single-group interventional pre-post design to assess the effect of an antioxidant-rich diet on Dietary Antioxidant Index (DAI) and metabolic syndrome risk.
  Participants will receive an antioxidant rich dietary intervention, and changes in DAI and metabolic syndrome parameters will be measured before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Antioxidant Index-Based Dietary Intervention Arm (Experimental): Participants in this arm will receive an antioxidant-rich dietary intervention designed to improve the Dietary Antioxidant Index (DAI). The intervention includes guidance to increase intake of fruits, vegetables, whole grains, legumes, and antioxidant-rich foods while limiting pro-oxidant and ultra-processed foods. Changes in DAI and metabolic syndrome components will be assessed before and after the intervention.
  Interventions: Other: Antioxidant-Focused Diet Intervention

INTERVENTIONS:
Other: Antioxidant-Focused Diet Intervention — This intervention specifically targets the Dietary Antioxidant Index (DAI) by increasing consumption of antioxidant-rich foods such as fruits, vegetables, whole grains, and legumes, while limiting pro-oxidant and ultra-processed foods. Unlike general healthy diet interventions, this study focuses on quantifiable antioxidant intake and its direct association with metabolic syndrome risk in urban adults.

SUMMARY:
Metabolic syndrome (MetS) is a cluster of metabolic disorders characterized by elevated levels of blood glucose, hypertension, dyslipidemia, and abdominal obesity. Globally, it is a major public health concern. International studies have linked higher Dietary Antioxidant Index with reduced risk of MetS, as antioxidants play a role in lowering the risk of MetS by reducing oxidative stress, a key contributor to its pathophysiology. Exploring this link in Pakistan can provide valuable insights for dietary strategies to reduce the risk of MetS.

DETAILED DESCRIPTION:
Background: Metabolic syndrome (MetS) is a cluster of metabolic disorders characterized by elevated levels of blood glucose, hypertension, dyslipidemia, and abdominal obesity. Globally, it is a major public health concern. International studies have linked higher Dietary Antioxidant Index (DAI) scores with reduced risk of MetS, as antioxidants play a role in lowering the risk of MetS by reducing oxidative stress, a key contributor to its pathophysiology. Exploring this link in Pakistan can provide valuable insights for dietary strategies to reduce the risk of MetS.

Hypothesis: A dietary intervention aimed at improving Dietary Antioxidant Index (DAI) scores beneficially affects Metabolic Syndrome risk factors among urban adults at risk of developing Metabolic Syndrome.

Material and Methods: A single-group pre-post human interventional study will be conducted among at-risk urban adults identified through the NCEP ATP III and WHO criteria. Dietary recalls will be analyzed in NutriSurvey using the Pakistan Food Composition Table, and any missing nutrient values will be supplemented from the Indian Food Composition Table. Nutrient data will be used to calculate the Dietary Antioxidant Index (DAI). Individuals with low DAI will receive dietary intervention.

Statistical Analysis: Pre-post changes in DAI and MetS markers will be assessed using paired t-tests, and Pearson's correlation will determine their associations using SPSS 25.

Expected Outcomes: The intervention is expected to reduce key Metabolic Syndrome risk factors while increasing individuals' awareness and motivation to adopt healthier behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years
* Metabolic syndrome risk (abdominal obesity & elevated BP as per NCEP ATP III criteria).
* Low fruit & veg intake (<5 serv./day) as per WHO.
* Willing to follow an intervention
* Non-pregnant or lactating
* Not diagnosed with malabsorption syndrome or chronic illness

Exclusion Criteria:

* Individuals < 18 years or > 45 years
* Not at risk of metabolic syndrome.
* Adequate intake of fruits & veg (≥ 5 serv./day) as per WHO
* Not willing
* Pregnant or lactating
* Diagnosed with malabsorption syndrome or chronic illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in Dietary Antioxidant Index (DAI) | Baseline and after 12 weeks of intervention
  DAI will be calculated from 24-hour dietary recalls to quantify total antioxidant intake. The primary objective is to assess whether the antioxidant-rich diet increases DAI in participants.
Change in Metabolic Syndrome Risk Score | Baseline and after 12 weeks of intervention
  A composite metabolic syndrome risk score will be calculated by summing standardized z-scores of waist circumference (cm), fasting blood glucose (mg/dL), systolic blood pressure (mmHg), triglycerides (mg/dL), and inversely weighted HDL-cholesterol (mg/dL) to generate a single continuous measure of overall metabolic syndrome risk.

SECONDARY OUTCOMES:
Change in Body Composition | Baseline and after 12 weeks of intervention
  Body composition, including body fat percentage and skeletal muscle mass, will be assessed using InBody analyzer to evaluate changes in body composition.

CONTACTS AND LOCATIONS:
Overall Officials: Qaisar Raza, Ph.D, Principal Investigator — UNIVERSITY OF VETERINARY & ANIMAL SCIENCES, LAHORE PAKISTAN.
Locations (1):
- University of Veterinary & Animal Sciences, Lahore Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No